CLINICAL TRIAL: NCT03968991
Title: VISIODOL: Validation of the VISIODOL® Scale for Screening of Pain in People With Visual Impairment
Brief Title: VISIODOL: Validation of the VISIODOL® Scale
Acronym: VISIODOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruits
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2018 PICKERING 2; 2018-A03370-55 (Other: 2018-A03370-55)
Record Dates: First submitted 2019-04-29; First posted 2019-05-31 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-01

CONDITIONS: Visual Deficiency; Congenital Blindness; Acquired Blindness
Keywords: Blinded population; Pain evaluation; Diagnostic tool
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteer group (Active Comparator): male or female healthy volunteers
  Interventions: Diagnostic Test: VISIODOL® (Diagnostic tool)
- Subjects with acquired visual impairment (Experimental): visual acquired disability
  Interventions: Diagnostic Test: VISIODOL® (Diagnostic tool)
- Subjects with congenital visual impairment (Experimental): Visual congenital disability
  Interventions: Diagnostic Test: VISIODOL® (Diagnostic tool)

INTERVENTIONS:
Diagnostic Test: VISIODOL® (Diagnostic tool) — Tool for assessing pain in the blind subject (with congenital or acquired deficiency)

SUMMARY:
The aim of this study is to validate the VISIODOL® scale for screening of pain in people with visual impairment.

DETAILED DESCRIPTION:
The VISIODOL® monocentric study conducted at Clermont-Ferrand University Hospital is a cross-disciplinary diagnostic tool validation performed in patients with acquired or congenital visual impairment and healthy sighted volunteers. Different evaluations by thermal (Pathway Médoc®) and mechanical (electronic Von Frey®) tests will allow to compare the new VISIODOL® scale with the numerical scale, which is a commonly used tool. The ergonomic quality, the satisfaction of use and the quality of life, stress, anxiety and catastrophism of the patients will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Subjects aged over 18 / under 60
* Male or female
* Subjects fasting from coffee, tea, Coca-Cola and others stimulants
* Sufficient understanding and cooperation to comply with the study requirements
* Agreed to provide written consent
* Affiliated to the social security
* Subjects with visual impairment (congenital or acquired)
* Subjects with no visual impairment (healthy group)

Exclusion Criteria:

* Subjects under 18 years old
* Administrative and legal criteria (tutorship, curatorship, without social security, in exclusion period of another study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using thermal tests. | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for different pain temperatures by hot thermal tests. The rating of the NS and VISIODOL® scales can range from 0 to 10.

SECONDARY OUTCOMES:
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using thermal tests. | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for sensitive threshold by hot thermal tests. The rating of the NS and VISIODOL® scales can range from 0 to 10.
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using thermal tests . | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for sensitive threshold by cold thermal tests. The rating of the NS and VISIODOL® scales can range from 0 to 10.
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using thermal tests. | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for pain threshold by cold thermal tests. The rating of the NS and VISIODOL® scales can range from 0 to 10.
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using mechanical tests. | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for sensitive threshold by electronic Von Frey®. The rating of the NS and VISIODOL® scales can range from 0 to 10.
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using mechanical tests. | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for pain threshold by electronic Von Frey. The rating of the NS and VISIODOL® scales can range from 0 to 10.
Validation of the VISIODOL® scale in screening of pain in people with visual impairment using the correlation coefficient between the intensities measured with the Numerical Scale (NS) and the VISIODOL® scale obtained by using mechanical tests. | Day 0 + 2 hours
  Determination of the correlation coefficient between NS and VISIODOL® scale for tolerance threshold by electronic Von Frey. The rating of the NS and VISIODOL® scales can range from 0 to 10.
Comparison of pain perception between the 3 groups | Day 0 + 1 hour
  comparison of NS and VISIODOL® scoring for pain threshold by hot thermal tests (Pathway Medoc®).
Evaluation of the ergonomic qualities of the scale | Day 0 + 1 hour
  ergonomic survey : Different ergonomic parameters such as length, width and granulometry will be evaluated using a questionnaire.
Evaluation of satisfaction of the use of the scale | Day 0 + 1 hour
  satisfaction survey : The satisfaction of the participants in the study will be collected by means of a questionnaire.
Evaluation of anxiety | Day 0 + 1 hour
  Hospital and Anxiety Depression Scale (HAD) : The Hospital Anxiety and Depression scale is a self-administered questionnaire in 14 items completed by the patient. It is used to determine the levels of anxiety and depression. Seven of the items relate to anxiety and seven relate to depression. Global score ranges from 0 to 42.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Morel V, Goubayon J, Touron A, Leray V, Pereira B. A tactile pain evaluation scale for persons with visual deficiencies. Pain Med. 2023 Jul 5;24(7):855-861. doi: 10.1093/pm/pnad013. PMID 36809402